CLINICAL TRIAL: NCT01330472
Title: An Open Label, Randomized, Single Dose, Crossover Pivotal Bioequivalence Study Of Xanax XR Tablet 3 mg (Sourced From Caguas) Versus Xanax XR Tablet 3 mg (Sourced From Barceloneta) In Healthy Subjects
Brief Title: An Bioequivalence Study Of Xanax Extended Release Tablets From Two Different Manufacturing Sites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131025
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy Subjects
Keywords: Alprazolam; Xanax; Bioequivalence; Panic disorder with or without agoraphobia.
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xanax XR tablets 3 mg (sourced from Caugus) (Active Comparator): Xanax XR tablets 3 mg (sourced from Caugus), 1 x 3 mg (REFERENCE)
  Interventions: Drug: Xanax XR tablets 3 mg (sourced from Caugus)
- Xanax XR tablets 3 mg (sourced from Barceloneta), (Experimental): Xanax XR tablets 3 mg (sourced from Barceloneta), 1 x 3 mg (TEST)
  Interventions: Drug: Xanax XR tablets 3 mg (sourced from Barceloneta)

INTERVENTIONS:
Drug: Xanax XR tablets 3 mg (sourced from Caugus) — Tablets, 3 mg, single dose
  Arms: Xanax XR tablets 3 mg (sourced from Caugus)
Drug: Xanax XR tablets 3 mg (sourced from Barceloneta) — Tablets, 3 mg, single dose
  Arms: Xanax XR tablets 3 mg (sourced from Barceloneta),

SUMMARY:
Study to evaluate if Xanax sustained release tablets manufactured at two different sites provide similar drug levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 20 and 55 years, inclusive.
* An informed consent document signed and dated by the subject.

Exclusion Criteria:

* Evidence or history of clinically significant abnormality.
* A positive urine drug screen.
* Subjects who are hypersensitive to alprazolam or related compounds.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to infinity (AUCinf) of alprazolam | Predose, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose
Peak plasma conc (Cmax) of alprazolam | Predose, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose

SECONDARY OUTCOMES:
Area under the curve from zero to the last time point (AUClast) of alprazolam | Predose, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose
Area under the curve extrapolated (AUC%extrap) of alprazolam | Predose, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose
Terminal half life of alprazolam | Predose, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose
Time to peak concentration (Tmax) of alprazolam | Predose, and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131025&StudyName=An%20Bioequivalence%20Study%20Of%20Xanax%20Extended%20Release%20Tablets%20From%20Two%20Different%20Manufacturing%20Sites